| Home-based or traditional class HIIT in overweight women: effects on physical activity, body composition and cardiorespiratory fitness. A 3-arm randomized control trial |
|---|
| Ethics Comission for Scientific Investigation in Human Health and Well-being of Evora University approval number 21016 |
| 22 February 2021 |

## **Informed Consent**



The present study, carried out within the scope of the PhD thesis in Human Motricity at the University of Évora by doctoral student João Carmo, with the theme "HIIT training at home in overweight women - a randomized study with 3 groups", which aims to verify the effect of HIIT training in the context of the home and in the context of formal class.

This study is under the supervision of Jorge Bravo, PhD, Jorge Mota, PhD, and Armando Raimundo, PhD, declares that:

- Anonymity and confidentiality of your data will be maintained, as we enshrine professional secrecy as an obligation and a duty.

According to the above:

- I declare that all procedures relating to the ongoing investigation were clear and answered satisfactorily to all my questions;
- I understand that I have the right to ask, now and in the development of the study, any question about the study and the methods to be used;
- I understand the conditions and procedures, advantages and risks of participating in this study.
- They assured me that the files that concern the study will be kept confidential and that no information will be published or communicated, jeopardizing my privacy and identity;
- I understand that I am free to abandon the study at any time. After duly informed, I authorize participation in this study.

| Date://20 | |
|---------------|-----------------------|
| Participant | |
| | Documento of identity |
| Investigator: | |
| Signature: | |